CLINICAL TRIAL: NCT01807052
Title: Observational - Tissue Factor Expression in Bone Sarcomas
Brief Title: Biomarker Expression in Tissue Samples From Patients With Bone Sarcomas
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AOST10B2; NCI-2013-00112 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-AOST10B2 (Other: Children's Oncology Group)
Record Dates: First submitted 2013-03-06; First posted 2013-03-08 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Localized Osteosarcoma; Metastatic Osteosarcoma; Recurrent Osteosarcoma
MeSH Terms: conditions — Osteosarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: Tissue samples are analyzed for tumor factor expression levels by immunohistochemistry.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This trial studies biomarker expression in tissue samples from patients with bone sarcomas. Studying biomarker in tissue samples from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer

DETAILED DESCRIPTION:
STUDY SUBTYPE: Ancillary/Correlative

OBSERVATIONAL STUDY MODEL: Case-only

TIME PERSPECTIVE: Retrospective

BIOSPECIMEN RETENTION: Samples without DNA

BIOSPECIMEN DESCRIPTION: Tissue samples obtained from Cooperative Human Tissue Network (CHTN)

STUDY POPULATION DESCRIPTION: Patients enrolled on P9754 and AOST0121 clinical trials

SAMPLING METHOD: Non-probability sample

PRIMARY OBJECTIVES:

I. To determine if there is differential expression of tumor factor (TF) among patients with osteosarcoma.

II. To determine if there is an association between overall survival and disease free survival and the extent of TF expression.

III. To determine if TF expression correlates with presence of gross metastatic disease at presentation, and development of subsequent metastases.

OUTLINE:

Tissue samples are analyzed for tumor factor expression levels by immunohistochemistry.

ELIGIBILITY:
Inclusion Criteria:

* Tissue samples from patients with osteosarcomas obtained from the CHTN:

  * P9754 clinical trial for patients with non-metastatic osteosarcoma
  * AOST0121 clinical trial for patients with metastatic or recurrent osteosarcoma

Max Age: 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Tissue samples from patients with osteosarcomas obtained from the CHTN that participated in either study P9754 clinical trial for patients with non-metastatic osteosarcoma or AOST0121 clinical trial for patients with metastatic or recurrent osteosarcoma
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2009-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of high TF expression | 1 month
  Estimated in the analytic population as the number of samples in the population in which such expression is noted divided by 33. An assessment of the precision of such estimates will be provided by an exact binomial confidence interval. Comparison of normalized TF expression in non-metastatic versus metastatic patients will be done using the two-sample t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ranalli, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States